CLINICAL TRIAL: NCT05733975
Title: Decision Making Support for Parents and Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00111995; K23NS116453 (NIH)
Record Dates: First submitted 2023-01-24; First posted 2023-02-17 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Neonatal Critical Illness; Pediatric Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Critically Ill Infants (Other): Parent(s) of critically ill infants received the decision making guide intervention and could choose to share their completed tool with their infant's clinicians.
  Interventions: Other: Decision Making Guide
- Parent(s) of Critically Ill Infant (Other): Parent(s) of critically ill infants received the decision making guide intervention and could choose to share their completed tool with their infant's clinicians.
  Interventions: Other: Decision Making Guide
- Clinicians (Other): Parent(s) of critically ill infants received the decision making guide intervention and could choose to share their completed tool with their infant's clinicians.
  Interventions: Other: Decision Making Guide

INTERVENTIONS:
Other: Decision Making Guide — The tool includes a brief introduction to the tool and decision-making, a values clarification exercise, and a question prompt list.

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of a tool to support decision making for parents of critically ill infants.

DETAILED DESCRIPTION:
In this single-arm mixed methods prospective feasibility study, we will enroll infants, parents, and clinicians. The intervention is a paper-based decision guide that contains a values clarification exercise and question prompt list.

ELIGIBILITY:
Study participants will include English-speaking parents of critically ill infants and children admitted to Duke University Hospital.

Infant inclusion criteria will include

1. age < 1 year,
2. admission to a critical care unit, and
3. an anticipated serious health care decision

All parents of eligible infants will be considered for inclusion. Parent exclusion criteria will include 1) age < 18 years, 2) hearing or speech impairment, and 3) non-English speakers.

All clinicians of eligible infants will be considered for inclusion.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Lemmon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant level data

REFERENCES:
- [Background] Lemmon ME, Boss RD, Bonifacio SL, Foster-Barber A, Barkovich AJ, Glass HC. Characterization of Death in Neonatal Encephalopathy in the Hypothermia Era. J Child Neurol. 2017 Mar;32(4):360-365. doi: 10.1177/0883073816681904. Epub 2016 Dec 20. PMID 28193115
- [Background] Emanuel EJ, Emanuel LL. Four models of the physician-patient relationship. JAMA. 1992 Apr 22-29;267(16):2221-6. No abstract available. PMID 1556799
- [Background] Carlet J, Thijs LG, Antonelli M, Cassell J, Cox P, Hill N, Hinds C, Pimentel JM, Reinhart K, Thompson BT. Challenges in end-of-life care in the ICU. Statement of the 5th International Consensus Conference in Critical Care: Brussels, Belgium, April 2003. Intensive Care Med. 2004 May;30(5):770-84. doi: 10.1007/s00134-004-2241-5. Epub 2004 Apr 20. PMID 15098087
- [Background] White DB, Braddock CH 3rd, Bereknyei S, Curtis JR. Toward shared decision making at the end of life in intensive care units: opportunities for improvement. Arch Intern Med. 2007 Mar 12;167(5):461-7. doi: 10.1001/archinte.167.5.461. PMID 17353493
- [Background] Azoulay E, Chevret S, Leleu G, Pochard F, Barboteu M, Adrie C, Canoui P, Le Gall JR, Schlemmer B. Half the families of intensive care unit patients experience inadequate communication with physicians. Crit Care Med. 2000 Aug;28(8):3044-9. doi: 10.1097/00003246-200008000-00061. PMID 10966293
- [Background] Curtis JR, Engelberg RA, Wenrich MD, Shannon SE, Treece PD, Rubenfeld GD. Missed opportunities during family conferences about end-of-life care in the intensive care unit. Am J Respir Crit Care Med. 2005 Apr 15;171(8):844-9. doi: 10.1164/rccm.200409-1267OC. Epub 2005 Jan 7. PMID 15640361
- [Background] Cox CE, Lewis CL, Hanson LC, Hough CL, Kahn JM, White DB, Song MK, Tulsky JA, Carson SS. Development and pilot testing of a decision aid for surrogates of patients with prolonged mechanical ventilation. Crit Care Med. 2012 Aug;40(8):2327-34. doi: 10.1097/CCM.0b013e3182536a63. PMID 22635048
- [Background] Stacey D, Legare F, Lewis K, Barry MJ, Bennett CL, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2017 Apr 12;4(4):CD001431. doi: 10.1002/14651858.CD001431.pub5. PMID 28402085
- [Background] Cox CE, White DB, Hough CL, Jones DM, Kahn JM, Olsen MK, Lewis CL, Hanson LC, Carson SS. Effects of a Personalized Web-Based Decision Aid for Surrogate Decision Makers of Patients With Prolonged Mechanical Ventilation: A Randomized Clinical Trial. Ann Intern Med. 2019 Mar 5;170(5):285-297. doi: 10.7326/M18-2335. Epub 2019 Jan 29. PMID 30690645
- [Background] Boss RD, Hutton N, Sulpar LJ, West AM, Donohue PK. Values parents apply to decision-making regarding delivery room resuscitation for high-risk newborns. Pediatrics. 2008 Sep;122(3):583-9. doi: 10.1542/peds.2007-1972. PMID 18762529
- [Background] Zupancic JA, Kirpalani H, Barrett J, Stewart S, Gafni A, Streiner D, Beecroft ML, Smith P. Characterising doctor-parent communication in counselling for impending preterm delivery. Arch Dis Child Fetal Neonatal Ed. 2002 Sep;87(2):F113-7. doi: 10.1136/fn.87.2.f113. PMID 12193517
- [Derived] Lemmon ME, Bansal S, Nanduri N, Davalos A, Glass HC, Lord B, Moline K, Pilon B, Sharpe R, Brandon D, Hong H, Samsa G, Cox CE, Pollak KI. Feasibility of an Intervention to Support Shared Decision-Making for Critically Ill Infants. J Pediatr. 2025 Aug;283:114632. doi: 10.1016/j.jpeds.2025.114632. Epub 2025 May 2. PMID 40319938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on assessment of infant eligibility and approval from primary physician. Parental consent was obtained based on eligible participants. The first participant was enrolled on May 2, 2023 and the last participant was enrolled January 29, 2024.
Period: Overall Study
Arm/Group | Critically Ill Infants | Parent(s) of Critically Ill Infant | Clinicians
Started | 30 | 44 | 30
Completed | 30 | 42 | 30
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Measure Analysis Population Description: Demographic information includes 30 infants, 43 parents and 30 clinicians that completed demographic surveys. One parent was not included in this data due to withdrawal of participation before any data collection.
Groups:
- Total: Total of all reporting groups
Arm/Group | Critically Ill Infants | Parent(s) of Critically Ill Infant | Clinicians | Total
Number analyzed (Participants) | 30 | 43 | 30 | 103
Age, Continuous [Median (Inter-Quartile Range); unit: days] — Population: This row includes the infant population only. Infant age at enrollment is reported in days. Adults are not reported in this section.
  days
    Age at enrollment: number analyzed (Participants) | 30 | 0 | 0 | 30
    Age at enrollment | 20 [1.0 to 340.0] |  |  | 20 [1.0 to 340.0]
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: This row includes the adult population only (parents and clinicians). Infants are not reported in this section.
  years
    number analyzed (Participants) | 0 | 43 | 30 | 73
    (all) |  | 30.0 [19.0 to 41.0] | 41.0 [26.0 to 63.0] | 34.0 [19.0 to 63.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 30 | 22 | 62
  Male | 20 | 13 | 8 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 2 | 10
  Not Hispanic or Latino | 26 | 39 | 28 | 93
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 15 | 3 | 33
  White | 13 | 19 | 25 | 57
  More than one race | 1 | 4 | 0 | 5
  Unknown or Not Reported | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate (Critically Ill Infants)
Description: Intervention and study procedures considered feasible if infant enrollment rate is greater than or equal to 50%.
Time Frame: At enrollment (approximately 9 months)
Population: Eligible critically ill infants.
Measure: Count of Participants; unit: Participants
Arm/Group | Critically Ill Infants
Number analyzed (Participants) | 54
Participants
  Not enrolled/ consented | 24
  Enrolled/ Consented | 30

2. Primary Outcome: Complete Data Collection (Critically Ill Infants)
Description: Complete data collection defined as all eligible infant, parent, and clinician data points collected for a given case and was determined at the level of the critically ill infant. Data points for which the participant withdrew prior to relevant data collection were excluded. Intervention and study procedures considered feasible if complete data collection rate is greater than or equal to 80%.
Time Frame: approximately 9 months
Population: Critically ill infants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Critically Ill Infants
Number analyzed (Participants) | 30
Participants
  Completed data collection | 29
  Incomplete data collection | 1

3. Secondary Outcome: Parent and Clinician Acceptability
Description: Acceptability will be measured using an acceptability questionnaire, consisting of close-ended items with 5-point likert scale response options (strongly disagree, disagree, neither agree or disagree, agree, strongly agree).
Time Frame: Up to 4 weeks following use of the tool
Population: Not applicable to the infant group.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent(s) of Critically Ill Infant | Clinicians
Number analyzed (Participants) | 40 | 30
Participants
  Found to be helpful (agreed/strongly agreed) | 30 | 28
  Found to be helpful (all other response items) | 10 | 2
  Would recommend to other parents (agreed/ Strongly agreed) | 35 | 29
  Would recommend to other parents (all other response items) | 5 | 1
  Would use in the future (agreed/strongly agreed) | 33 | 29
  Would use in the future (all other response items) | 7 | 1

4. Secondary Outcome: Parent Psychological Distress, as Measured by the Patient-Reported Outcomes Measurement Information System (PROMIS)
Description: PROMIS measures assess the extent to which patients experience challenges with symptoms over the past 7 days. Scores are derived using a standardized T-score metric, with a mean of 50 and a standard deviation of 10. Higher scores reflect greater symptom severity.
Time Frame: Baseline, and up to 4 weeks following use of the tool
Population: Only applicable to the parent group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Parent(s) of Critically Ill Infant
Number analyzed (Participants) | 41
score on a scale
  Baseline PROMIS: Ability to Participate in Social Roles and Activities | 53.8 [44.2 to 64.2]
  Post Intervention PROMIS: Ability to Participate in Social Roles and Activities: number analyzed (Participants) | 40
  Post Intervention PROMIS: Ability to Participate in Social Roles and Activities | 51.8 [44.2 to 64.2]
  Baseline PROMIS: Emotional Distress-Anxiety | 57.7 [51.3 to 64.9]
  Post Intervention PROMIS: Emotional Distress-Anxiety: number analyzed (Participants) | 40
  Post Intervention PROMIS: Emotional Distress-Anxiety | 57.5 [48.9 to 62.7]
  Baseline PROMIS: Emotional Distress - Depression | 47.8 [38.2 to 55.1]
  Post Intervention PROMIS: Emotional Distress - Depression: number analyzed (Participants) | 40
  Post Intervention PROMIS: Emotional Distress - Depression | 52.5 [42.9 to 55.8]
  Baseline PROMIS: Fatigue | 53.9 [48.6 to 58.9]
  Post Intervention: Fatigue: number analyzed (Participants) | 40
  Post Intervention: Fatigue | 53.2 [46.4 to 62.4]
  Baseline PROMIS: Pain Interference | 49.2 [41.6 to 55.7]
  Post Intervention PROMIS: Pain Interference: number analyzed (Participants) | 40
  Post Intervention PROMIS: Pain Interference | 41.6 [41.6 to 51.9]
  Baseline PROMIS: Physical Function | 57.0 [47.8 to 57.0]
  Post Intervention PROMIS: Physical Function: number analyzed (Participants) | 40
  Post Intervention PROMIS: Physical Function | 57.0 [47.3 to 57.0]
  Baseline PROMIS: Sleep Disturbance | 50.1 [49.0 to 57.7]
  Post-Intervention PROMIS: Sleep Disturbance: number analyzed (Participants) | 40
  Post-Intervention PROMIS: Sleep Disturbance | 51.4 [47.0 to 56.3]

5. Secondary Outcome: Parent Preparation for Decision Making, as Measured by the PrepDM
Description: Items can be summed and scored. Score ranges from 0-100, where a higher score indicates higher perceived preparedness for decision making.
Time Frame: Up to 4 weeks following use of the tool
Population: Only applicable to the parent group.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Parent(s) of Critically Ill Infant
Number analyzed (Participants) | 40
score on a scale | 73.75 [59.38 to 90.00]

ADVERSE EVENTS:
Time Frame: Up to 4 weeks following use of the tool
Arm/Group | Critically Ill Infants | Parent(s) of Critically Ill Infant | Clinicians
All-Cause Mortality (participants affected / at risk) | 4/30 | 0/44 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/44 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/44 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT05733975/Prot_001.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT05733975/SAP_002.pdf
  • Informed Consent Form (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT05733975/ICF_000.pdf